CLINICAL TRIAL: NCT03550001
Title: Prospective Randomized Clinical Trial of Carbon Nanoparticles as Lymph Node Tracer in Rectal Cancer After Neoadjuvant Radiochemotherapy
Brief Title: Carbon Nanoparticles as Lymph Node Tracer in Rectal Cancer After Neoadjuvant Radiochemotherapy
Acronym: CALOR-NAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: YE Yingjiang (Other)
Responsible Party: Sponsor-Investigator, YE Yingjiang, Professor of Surgery, Director of Department of Gastroenterological Surgery, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-PKUPH077
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Rectal Cancer
Keywords: locally advanced rectal cancer; lymph node yeild; lymph node tracer; stage shift; prognosis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection CNP before NAT (Experimental): Inject carbon nanoparticle as a lymph node tracer before the patient receive neoadjuvant therapy.
  Interventions: Procedure: Injection CNP before NAT
- No injection (No Intervention): Do not inject carbon nanoparticle during the treatment.

INTERVENTIONS:
Procedure: Injection CNP before NAT — Injection carbon nanoparticle via rectal mucosa before neoadjuvant therapy
  Arms: Injection CNP before NAT

SUMMARY:
The purpose of this study is to evaluate whether injection of carbon nanoparticle as a lymph node tracer before neoadjuvant radiochemotherapy in rectal cancer can increase lymph node yield after surgery compared which do not inject.

DETAILED DESCRIPTION:
This is the randomized controlled, multi-centers，and open-labeled study. The lymph node yield was significantly decreased in rectal cancer after neoadjuvant radiochemotherapy (NAT), hard for pathologists to detect, and is difficult to meet the guideline that minimun of 12 lymph nodes should be retrived after surgery in colorectal cancer. Carbon nanoparticle (CNP) is a specific lymph node tracer, which only dyeing the lymph node, and can keep the lymph node in dyeing state in at least half year. The inverstigator attempted to compare the amount of lymph node yield after surgery in locally advanced rectal caner between injection CNP before NAT and no injection CNP before NAT. In this study, the participants with clinical TNM stage T3+ or N+ will be recruited. The participants will be randomized (1:1 ratio) to a control and intervention arm. The participants in the control arm will not receive injection of any kind lymph node tracers. The participants in the intervention arm will receive injection of CNP before NAT. And the specimen would be evaluated by the pathologist.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Histologically confirmed adenocarcinoma;
3. The rectal adenocarcinoma 0-12cm from the anal margin;
4. Clinical TNM stage: T3+ or N+;
5. Untreated patients (who have not received treatment including radiotherapy, chemotherapy, and surgery);
6. Good liver and kidney function, without contraindications for radiotherapy, chemotherapy or surgery;
7. Able and willing to give informed consent to participate;

Exclusion Criteria:

1. Malignant tumor history or other malignant tumors;
2. Emergency operations such as intestinal obstruction, perforation and hemorrhage;
3. Pregnant or lactating women;
4. History of severe mental illness;
5. Contraindications for radiotherapy, chemotherapy and surgery;
6. Conditions that the researcher thinks it is not suitable for selection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
lymph node yield | up to 30days after total mesorectal excision
  Amount of lymph node yield, dyeing lymph node, positive lymph node and the dyeing positive lymph node

SECONDARY OUTCOMES:
Impact on surgical operations | Time of surgery
  The impact of CNP to operational level
Quality of surgery | Time of surgery
  Quality of surgery determined using the mesorectal grading system
Surgery morbidity | 30 days and 12-months
  Surgical morbidity reported according to Clavien-Dindo classification
Overall survival | 5-years
  Overall Survival is defined as the time from the date of surgery to the date of death
Disease free survival | 5-years
  Disease Free Survival is defined as the time from the date of surgery to the date of the local recurrence, and/or distant disease, or tumor-related death
Local recurrence rate | 5-years
  Local recurrence rate is defined as the time from the date of surgery to the date of the local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Yingjiang Ye, MD,PhD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided
We need to discuss with other centers, then decide whether to share IPD

REFERENCES:
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Background] Mechera R, Schuster T, Rosenberg R, Speich B. Lymph node yield after rectal resection in patients treated with neoadjuvant radiation for rectal cancer: A systematic review and meta-analysis. Eur J Cancer. 2017 Feb;72:84-94. doi: 10.1016/j.ejca.2016.10.031. Epub 2016 Dec 24. PMID 28027520
- [Background] Gurawalia J, Dev K, Nayak SP, Kurpad V, Pandey A. Less than 12 lymph nodes in the surgical specimen after neoadjuvant chemo-radiotherapy: an indicator of tumor regression in locally advanced rectal cancer? J Gastrointest Oncol. 2016 Dec;7(6):946-957. doi: 10.21037/jgo.2016.09.03. PMID 28078118
- [Background] Kim HJ, Jo JS, Lee SY, Kim CH, Kim YJ, Kim HR. Low Lymph Node Retrieval After Preoperative Chemoradiation for Rectal Cancer is Associated with Improved Prognosis in Patients with a Good Tumor Response. Ann Surg Oncol. 2015;22(6):2075-81. doi: 10.1245/s10434-014-4235-z. Epub 2014 Nov 14. PMID 25395150
- [Background] Xu Z, Berho ME, Becerra AZ, Aquina CT, Hensley BJ, Arsalanizadeh R, Noyes K, Monson JRT, Fleming FJ. Lymph node yield is an independent predictor of survival in rectal cancer regardless of receipt of neoadjuvant therapy. J Clin Pathol. 2017 Jul;70(7):584-592. doi: 10.1136/jclinpath-2016-203995. Epub 2016 Dec 8. PMID 27932667
- [Background] Lykke J, Jess P, Roikjaer O; Danish Colorectal Cancer Group. A minimum yield of twelve lymph nodes in rectal cancer remains valid in the era of neo-adjuvant treatment : results from a national cohort study. Int J Colorectal Dis. 2015 Mar;30(3):347-51. doi: 10.1007/s00384-015-2145-6. Epub 2015 Feb 5. PMID 25652878
- [Background] Lykke J, Jess P, Roikjaer O; Danish Colorectal Cancer Group. Increased Lymph Node Yield Is Associated With Improved Survival in Rectal Cancer Irrespective of Neoadjuvant Treatment: Results From a National Cohort Study. Dis Colon Rectum. 2015 Sep;58(9):823-30. doi: 10.1097/DCR.0000000000000429. PMID 26252843
- [Background] Bhangu A, Kiran RP, Brown G, Goldin R, Tekkis P. Establishing the optimum lymph node yield for diagnosis of stage III rectal cancer. Tech Coloproctol. 2014 Aug;18(8):709-17. doi: 10.1007/s10151-013-1114-8. Epub 2014 Feb 11. PMID 24515286
- [Background] Carvalho C, Glynne-Jones R. Challenges behind proving efficacy of adjuvant chemotherapy after preoperative chemoradiation for rectal cancer. Lancet Oncol. 2017 Jun;18(6):e354-e363. doi: 10.1016/S1470-2045(17)30346-7. PMID 28593861
- [Background] Horne J, Carr NJ, Bateman AC, Kandala N 2nd, Adams J, Silva S, Ryder I. A comparison of formalin and GEWF in fixation of colorectal carcinoma specimens: rates of lymph node retrieval and effect on TNM staging. J Clin Pathol. 2016 Jun;69(6):511-7. doi: 10.1136/jclinpath-2015-203281. Epub 2015 Nov 30. PMID 26621110
- [Background] Yegen G, Keskin M, Buyuk M, Kunduz E, Balik E, Saglam EK, Kapran Y, Asoglu O, Gulluoglu M. The effect of neoadjuvant therapy on the size, number, and distribution of mesorectal lymph nodes. Ann Diagn Pathol. 2016 Feb;20:29-35. doi: 10.1016/j.anndiagpath.2015.10.008. Epub 2015 Oct 29. PMID 26706785
- [Background] Munster M, Hanisch U, Tuffaha M, Kube R, Ptok H. Ex Vivo Intra-arterial Methylene Blue Injection in Rectal Cancer Specimens Increases the Lymph-Node Harvest, Especially After Preoperative Radiation. World J Surg. 2016 Feb;40(2):463-70. doi: 10.1007/s00268-015-3230-2. PMID 26310202
- [Background] Farinella E, Vigano L, Fava MC, Mineccia M, Bertolino F, Capussotti L. In vivo lymph node mapping and pattern of metastasis spread in locally advanced mid/low rectal cancer after neoadjuvant chemoradiotherapy. Int J Colorectal Dis. 2013 Nov;28(11):1523-9. doi: 10.1007/s00384-013-1727-4. Epub 2013 Jul 23. PMID 23877264
- [Background] Zhang XM, Liang JW, Wang Z, Kou JT, Zhou ZX. Effect of preoperative injection of carbon nanoparticle suspension on the outcomes of selected patients with mid-low rectal cancer. Chin J Cancer. 2016 Apr 4;35:33. doi: 10.1186/s40880-016-0097-z. PMID 27044280
- [Background] Wang Y, Deng H, Chen H, Liu H, Xue Q, Yan J, Li G. Preoperative Submucosal Injection of Carbon Nanoparticles Improves Lymph Node Staging Accuracy in Rectal Cancer after Neoadjuvant Chemoradiotherapy. J Am Coll Surg. 2015 Nov;221(5):923-30. doi: 10.1016/j.jamcollsurg.2015.07.455. Epub 2015 Aug 20. PMID 26362137
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Mandard AM, Dalibard F, Mandard JC, Marnay J, Henry-Amar M, Petiot JF, Roussel A, Jacob JH, Segol P, Samama G, et al. Pathologic assessment of tumor regression after preoperative chemoradiotherapy of esophageal carcinoma. Clinicopathologic correlations. Cancer. 1994 Jun 1;73(11):2680-6. doi: 10.1002/1097-0142(19940601)73:113.0.co;2-c. PMID 8194005